CLINICAL TRIAL: NCT04288947
Title: Changing the Culture of Disrespect and Abuse in Maternity Care in Kumasi, Ghana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kwame Nkrumah University of Science and Technology (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1K43TWO1122--01
Record Dates: First submitted 2020-02-18; First posted 2020-02-28 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2022-01

CONDITIONS: Behavior Problem
Keywords: Disrespect and Abuse; Childbirth; Maternity Care
MeSH Terms: conditions — Mental Disorders | interventions — Prenatal Care

STUDY DESIGN:
Intervention Model Description: Training of midwives on 4 respectful maternal care modules.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Usual Care (Other): Training of midwives on 4 respectful maternal care modules.
  Interventions: Other: Disrespect and Abuse in Maternity Care

INTERVENTIONS:
Other: Disrespect and Abuse in Maternity Care — Changing the culture of disrespect and abuse in maternity care

SUMMARY:
Using a public health facility Komfo Anokye Teaching Hospital in Ghana the overall goal of the research is to examine: 1) the feasibility of implementing respectful care modules (RMC-M) in Kumasi, Ghana; 2) whether exposure to RMC-M increases participants perception of respectful maternity care in a public hospital setting in Ghana; and 3) the efficacy of RMC-M in changing midwives' attitudes, behaviors and clinical practice patterns. To achieve Aim 1, qualitative and quantitative study designs will be used to assess for reliability of implementation, usefulness, and patient responsiveness. Based on data collected, feasibility will be examined and the RMC-M will be further modified as needed prior to beginning Aim 2. To achieve Aim 2, a two group study design will be used, with one group of midwives receiving training on the RMC- M and the other not receiving any training. Participants receiving care from these two groups of midwives will be followed through intrapartum and surveyed postpartum to examine their perceptions of the care they received. To achieve Aim 3, a pre-post study design will examine whether expose to a RMC-M changes midwives' attitudes, behaviors, and clinical care of participants during labor and delivery.

DETAILED DESCRIPTION:
There is a growing recognition of disrespectful and abusive care of pregnant women during labor and delivery. Fear of maltreatment during labor and delivery has been identified as one barrier that prevents pregnant women from delivering in a facility.[1-3]. Pregnant Women report lack of sympathy and empathy, neglect, rudeness and verbally abusive behaviour, physically abusive behavior, lack of temperamental control, inadequate attention, and lack of privacy in skilled health care centres.[3,4] These form barriers to effective use of facilities[3,5,6] for childbirth as pregnant women recount that they receive better health care at home than in health facilities which is the only setting where skilled birth is provided in Ghana. Additionally, facility-based childbirth is known to avert mortality associated with deliveries which are often not detectable during prenatal care.[5,6] Currently, 1500 women die daily in sub-Saharan Africa from complications related to childbirth. [7,8] In the developing world, the life-time hazard of a woman dying from risks associated with pregnancy and child-birth is more than 300 times greater than for a woman living in a developed country; no other mortality rate has this disparity.[9] In Ghana, the current maternal mortality ratio is 380 per 100,000 live births and only 42% of women receive skilled childbirth care.

Four Respectful Maternity Care Modules (RMC-M) were developed from data collected during the candidate's dissertation research on disrespect and abuse in intrapartum care at four public hospitals in Ghana and from literature on the state of the science on disrespect and abuse. The content for four evidence-based modules includes topics on: 1) respect and dignity in childbirth; 2) communication; 3) focused antenatal care; and 4) use of alternative birthing positions for delivery. The modules use interactive teaching and learning methods such as role play, discussion, brain-storming, demonstration, and case study to discover acceptable practices, skills, and attitudes for respectful care provision. The intervention has the potential to improve pregnant women's experience of facility-based childbirth, therefore increasing satisfaction and decreasing home delivery. The RMC-M is proposed for midwives working in prenatal, intrapartum and postnatal facility-based childbirth units. Despite the proposed strengths of the RMC-M as a tool to improve perceptions of maternity care with facility-based childbirth, the fidelity and uptake of the intervention have not been tested. The purpose of this study is to test an intervention to promote respectful facility-based maternity care that can be delivered by midwives in Ghana in a public hospital setting through the following specific aims:

Specific Aim #1: Examine the feasibility of implementing respectful maternity care modules in Kumasi, Ghana.

The investigators will assign 10 professional midwives to receive training on Respectful Maternity Care Modules (RMC-M). During the training, we will use qualitative and quantitative analytic techniques to examine the feasibility of implementing the RMC-M in Ghana focused on: 1) reliability of implementation, 2) usefulness, and 3) patient responsiveness. Based on data collected, feasibility will be examined and the RMC-M will be further modified as needed prior to beginning Aim 2.

Specific Aim #2: Examine whether exposure to RMC-M increases Ghanaian women's perception of respectful maternity care in a public hospital setting in Ghana.

In order to meet aim #2, a two-group comparison design will be used with one group of pregnant women (n=62) receiving care from midwives trained in the RMC-M and the other group of pregnant women (n=62) receiving care from midwives who received a four module program in basic emergency obstetric and newborn care (BEmONC). Ten additional midwives will be trained in BEmONC prior to data collection. Data will be collected from postpartum women on their perception of intrapartum care.

It is hypothesized that postpartum women who receive care from midwives trained in the RMC-M interventions will score higher on a RMC scale than those women in the comparison group.

Specific Aim #3: Examine the efficacy of RMC-M in changing midwives' attitudes, behaviors, and clinical practice patterns.

Using a pre-post study design to examine whether exposure to the RMC-M changes midwives' attitudes, behaviors, and clinical practice in the care of women during labor and delivery. The investigators will survey midwives prior to implementing training on the RMC-M and following completion of aim #2.

It is hypothesized that midwives trained in the RMC-M interventions will have a significant change in attitudes, behaviors, and clinical practice than those midwives in the comparison group.

ELIGIBILITY:
Inclusion Criteria:

* Midwives providing childbirth care in the various units of Komfo Anokye Teaching Hospital (KATH)
* Patients receiving maternity care from Midwives Trained or untrained on Respectful Maternity care modules at KATH

Exclusion Criteria:

* Midwives working in other Hospitals apart from KATH
* Patients receiving care from other units apart from the maternity unit of KATH

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 110 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Respectful maternal care to women during childbirth as assessed by post natal women during a survey and interview. | Up to 42 months
  Women are respected during maternal care and childbirth

CONTACTS AND LOCATIONS:
Overall Officials: Peter Donkor, Study Director — Kwame Nkrumah University of Science and Technology; Jody Lori, PhD, Study Director — University of Michigan
Locations (1):
- Komfo Anokye Teaching Hospital, Kumasi, Ghana

IPD SHARING:
Plan to Share IPD: No